CLINICAL TRIAL: NCT04396301
Title: Effect of Intracameral Injection of Preservative Free, Fixed Concentration of Combined Mydriatic Plus Anaesthetic Formulation on Corneal Endothelial Cell Count in Phacoemulsification
Brief Title: Effect of Intracameral Injection of Mydriatic Plus Anaesthetic Combination on Corneal Endothelial Count in Phaco
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Elshewy, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CU-oph-02-2019
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Corneal Endothelial Cell Loss; Mydriasis; Cataract
Keywords: corneal endothelial cell count; Fydrane; mixed mydriatic and anaesthetic combination; intracameral mydriatic; mydriasis; phacoemulsification
MeSH Terms: conditions — Corneal Endothelial Cell Loss; Mydriasis; Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fydrane group (Active Comparator): Fydrane is injected intracamerally at the beginning of cataract surgery after the first incision, at a dose of 0.2 ml of solution, in only one injection. Fydrane®: (Manufacturer DELPHARM TOURS, FRANCE). No preoperative topical eye drops are used.
  Interventions: Drug: Fydrane®: (Manufacturer DELPHARM TOURS, FRANCE).
- Reference group: (No Intervention): not injected with intracameral Fydrane. Pupillary dilatation in this group is achieved using preoperative topical eye drops: cyclopentolate hydrochloride 1% and tropicamide 1 % one drop every 15 min for 1 hour preoperatively.

INTERVENTIONS:
Drug: Fydrane®: (Manufacturer DELPHARM TOURS, FRANCE). — Fydrane®. The active substances in Fydrane are: tropicamide 0.04 mg (anticholinergic), phenylephrine hydrochloride 0.62 mg (alpha sympathomimetic) and Lidocaine hydrochloride 2 mg (amide type local anaesthetics) for each 0.2 ml dose, equivalent to 0.2 mg of tropicamide, 3.1 mg of phenylephrine hydrochloride and 10 mg of lidocaine hydrochloride for 1 ml.
  Other Names: Mydrane
  Arms: Fydrane group

SUMMARY:
Study evaluates safety of intracameral injection of Fydrane (tropicamide 0.02%, phenylephrine 0.31% and lidocaine 1%) on corneal endothelium, and efficiency in maintaining pupillary dilatation during phacoemulsification surgery.

DETAILED DESCRIPTION:
in this prospective randomized controlled study, 30 eyes of 30 patients undergoing phacoemulsification with intraocular lens (IOL) implantation, were assigned into 2 groups. 15 eyes (Fydrane group) received 0.2ml of Fydrane just after the first incision. While 15 eyes (Reference group) received a topical regimen of one drop of each of cyclopentolate hydrochloride 1% and tropicamide 1 %, every 15 min for 1 hour preoperatively. The main outcome measures were safety on corneal endothelium, by comparing the preoperative and 3 weeks postoperative corneal endothelium cell count in the two groups. Efficacy was also evaluated by measuring pupil size using surgical caliper at certain timings during surgery: before capsulorhexis and before intraocular lens (IOL) implantation, in both groups.

ELIGIBILITY:
Inclusion Criteria:

* medium density cataract (nuclear II to III)

Exclusion Criteria:

* soft or hard density cataract (nuclear I or IV)
* history of ocular trauma or previous intraocular surgery
* iatrogenic, congenital or traumatic cataract
* associated eye disease e.g. pseudoexofoliation syndrome
* associated pre-existing corneal endothelial disease e.g. Fuchs dystrophy
* associated systemic disease that can affect endothelium,

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
safety of intracameral Fydrane on endothelial cell count | 3 weeks postoperative
  evaluates safety of Fydrane on corneal endothelium, assessed by calculating percentage of endothelial cell loss at 3 weeks postoperative

SECONDARY OUTCOMES:
effect of Fydrane on pupil diameter during phacoemulsification | pupil diameter is measured using surgical caliper at certain timings during surgery (before capsulorhexis and before IOL implantation)
  Fydrane Efficacy in achieving and maintaining mydiasis, is evaluated by measuring pupil diameter using surgical caliper at certain timings during surgery (before capsulorhexis and before IOL implantation)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University - Kasr Alainy hospital, Cairo, Egypt